CLINICAL TRIAL: NCT06033950
Title: A Randomized, Double-blind, Placebo-controlled Pragmatic Study to Evaluate Finerenone on Clinical Efficacy and Safety in Patients with Heart Failure and Reduced Ejection Fraction Who Are Intolerant of or Not Eligible for Treatment with Steroidal Mineralocorticoid Receptor Antagonists (FINALITY-HF)
Brief Title: A Study to Evaluate Finerenone on Clinical Efficacy and Safety in Patients with Heart Failure Who Are Intolerant or Not Eligible for Treatment with Steroidal Mineralocorticoid Receptor Antagonists
Acronym: FINALITY-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Collaborators: St. Luke's Hospital, Kansas City, Missouri (Other); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202304CPC
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Reduced ejection fraction; Symptomatic heart failure
MeSH Terms: conditions — Heart Failure | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Experimental)
  Interventions: Drug: Finerenone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — Oral finerenone.
  Arms: Finerenone
Drug: Placebo — Matching oral placebo.
  Arms: Placebo

SUMMARY:
Finerenone will be compared to placebo to determine efficacy and safety of treatment in patients with heart failure and reduced ejection fraction (HFrEF) who are intolerant or ineligible to receive treatment with steroidal mineralocorticoid receptor antagonists (sMRA).

DETAILED DESCRIPTION:
This is an international, randomized, double-blind, placebo-controlled trial of finerenone for the treatment of heart failure patients with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Provide electronic or written informed consent, either personally or through a legally authorized representative, as permitted by local regulations
* Age ≥18 years or legal age of majority if >18 years in the participant's country of residence
* Symptomatic HFrEF per protocol defined criteria
* Not on sMRA due to history of intolerance, contraindication, or ineligibility for treatment
* Negative pregnancy test and agreement to use adequate contraception during trial (female participants only)

Exclusion Criteria:

* Treatment with non-steroidal MRA (nsMRA)
* Documented prior history of severe hyperkalemia in the setting of MRA use
* eGFR < 25 mL/min/1.73m² and / or potassium > 5.0 mmol/L
* Acute myocardial infarction, coronary revascularization, valve replacement/repair, or implantation of a cardiac resynchronization therapy device within 30 days or planned
* Prior or planned heart transplant
* Hemodynamically significant (severe) uncorrected primary cardiac valvular disease considered by the investigator to be the primary cause of heart failure
* Symptomatic bradycardia or second- or third-degree heart block without a pacemaker
* Cardiomyopathy due to known acute inflammatory heart disease, infiltrative diseases, accumulation diseases, muscular dystrophies, cardiomyopathy with reversible causes, hypertrophic obstructive cardiomyopathy, complex congenital heart disease, or pericardial constriction
* Probable alternative cause of participant's HF
* Concomitant systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors, or moderate or potent CYP3A4 inducers
* Known hypersensitivity to the IP (active substance or excipients)
* Any other condition or therapy which would make the participant unsuitable for the study
* Concurrent or previous participation in another interventional clinical study using an investigational agent within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of cardiovascular (CV) death or HF event. | Ongoing, up to ~30 months
  - Time to first CV death or HF event with finerenone compared to placebo.
Number of serious adverse events | Ongoing, up to ~30 months
  - Serious adverse events (excluding efficacy endpoints) with finerenone compared to placebo.
Number of adverse events leading to discontinuation of study drug. | Ongoing, up to ~30 months
  - Number of adverse events leading to discontinuation of investigational product with finerenone compared to placebo.

SECONDARY OUTCOMES:
Timing and occurrence of total CV deaths and HF events | Ongoing, up to ~30 months
  - Timing and occurrence of total (first and subsequent) events of CV death and HF events and CV deaths with finerenone compared to placebo.
Timing and occurrence of total HF events | Ongoing, up to ~30 months
  Timing and occurrence of total (first and recurrent) HF events with finerenone compared to placebo.
Change in Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) from baseline to Month 6. | 180 days
  - Change in KCCQ-TSS with finerenone compared to placebo.
Time to CV death. | Ongoing, up to ~30 months
  - Time to CV death with finerenone compared to placebo.
Time to all-cause death. | Ongoing, up to ~30 months
  - Time to all-cause mortality with finerenone compared to placebo.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - FIN-10004 Fairhope, AL Investigational Site, Fairhope, Alabama
  - FIN-10075 San Diego, CA Investigational Site, San Diego, California
  - FIN-10002 Kansas City, MO Investigational Site, Kansas City, Missouri
  - FIN-10015 Austin, TX Investigational Site, Austin, Texas
- Brazil (3):
  - FIN-21003 Goiania, Goias Investigational Site, Goiânia, Goiás
  - FIN-21049 Sao Paulo, Investigational Site, Sao Paulp, Sap Paulo
  - FIN-21004 Braganca Paulista, Investigational Site, Bragança Paulista, São Paulo
- FIN-11012 Surrey, BC Investigational Site, Surrey, British Columbia, Canada